CLINICAL TRIAL: NCT00125905
Title: Effectiveness of a Stepped Primary Care Smoking Cessation Intervention Based on an Evidence Based Clinical Practice Guideline (ISTAPS Project)
Brief Title: ISTAPS: A Stepped Primary Care Smoking Cessation Intervention
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Fundacio d'Investigacio en Atencio Primaria Jordi Gol i Gurina (Other)
Collaborators: Preventive Services and Health Promotion Research Network (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PI021471; PI021471; G03/170
Record Dates: First submitted 2005-08-01; First posted 2005-08-02 (Estimated); Last update posted 2009-09-30 (Estimated); Status verified 2003-11

CONDITIONS: Smoking Cessation
Keywords: Primary Care; Smoking Cessation; Stages of Change Model; Health Education; Clinical Practice guideline
MeSH Terms: conditions — Smoking Cessation; Health Education | interventions — Counseling; Motivational Interviewing; Nicotine Chewing Gum; Transdermal Patch; Bupropion

INTERVENTIONS:
Behavioral: Advice
Behavioral: Motivational Interviewing
Drug: Nicotine Gum and Patch
Drug: Bupropion

SUMMARY:
Primary care centers can play a very important role in helping people to stop smoking. There is a large body of research on the effectiveness of specific interventions especially addressed to people who want to stop smoking. In addition to that, there are no studies with a large sample of individuals included that tested the complete range of interventions recommended nowadays for helping people in the different smoking cessation stages of change and with different degrees of physical and psychological dependence, especially including motivational interviewing in those not interested in cessation in the very next weeks. This study will test a complex intervention that at first classifies smokers in stages and after that treats every smoker according to what stage he/she is in at the moment, his/her degree of dependence and his/her own characteristics.

DETAILED DESCRIPTION:
OBJECTIVES:

* To evaluate the effectiveness of a stepped smoking cessation intervention based on a transtheoretical model of change that uses the pharmacological and no-pharmacological methods proposed by evidence based Clinical Practice Guidelines for smoking cessation from primary care centers.
* To assess the health status change in relationship with the smoking cessation process.

DESIGN: Cluster randomized clinical trial

Unit of Randomization: Care basic unit (family physician or nurse that cares for the same group of patients). Intention to treat analysis.

PARTICIPANTS: 2911 smokers (ages 14-75 years) consulting for any reason to primary care centers

INTERVENTION: 6-month implementation of recommendations of a Clinical Practice Guideline that includes motivational consulting for smokers at the precontemplation - contemplation stage; brief intervention for smokers in preparation-action who do not want help; intensive intervention with pharmacotherapies for smokers in preparation-action who want help; and reinforcing intervention in the maintenance stage.

CONTROL: Usual care

MEASUREMENT: Self reported abstinence confirmed by an expired air carbon monoxide concentration of 10 parts per millions or less; Point prevalence at the end of intervention, 1 and 2 years after the beginning of intervention; Continuous abstinence rate for 1 year; Change of stage in the smoking cessation process; Health status measured by SF-36.

ELIGIBILITY:
Inclusion Criteria:

* Smokers
* Accept participation and follow-up by phone interviews for 2 years

Exclusion Criteria:

* Terminal illness
* Active addictive behaviours or important health problems

Ages: 14 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 3012
Dates: Start 2003-10; Study Completion 2006-07

PRIMARY OUTCOMES:
Self reported abstinence confirmed by an expired air carbon monoxide concentration of 10 parts per millions or less
Point prevalence at the end of intervention, 1 and 2 years after the beginning of intervention
Continuous abstinence rate for 1 year
Change of stage in the smoking cessation process

SECONDARY OUTCOMES:
Health status measured by SF-36

CONTACTS AND LOCATIONS:
Overall Officials: Carmen Cabezas-Peña, MD, Principal Investigator — Jordi Gol I Gurina Foundation-ICS
Locations (1):
- Jordi Gol i Gurina Foundation-Primary Care Research Institute, Barcelona, Barcelona, Spain

REFERENCES:
- [Derived] Puente D, Cabezas C, Rodriguez-Blanco T, Fernandez-Alonso C, Cebrian T, Torrecilla M, Clemente L, Martin C; ISTAPS study group investigators. The role of gender in a smoking cessation intervention: a cluster randomized clinical trial. BMC Public Health. 2011 May 23;11:369. doi: 10.1186/1471-2458-11-369. PMID 21605389
- [Derived] Cabezas C, Advani M, Puente D, Rodriguez-Blanco T, Martin C; ISTAPS Study Group. Effectiveness of a stepped primary care smoking cessation intervention: cluster randomized clinical trial (ISTAPS study). Addiction. 2011 Sep;106(9):1696-706. doi: 10.1111/j.1360-0443.2011.03491.x. Epub 2011 Jul 22. PMID 21561497